CLINICAL TRIAL: NCT02792049
Title: Single Rescuer Ventilation Using a Bag Valve Mask With Integrated Internal Handle Versus Standard Bag Valve Mask in a Manikin Model: A Randomized Crossover Trial
Brief Title: Ventilation Using a Bag Valve Mask With Integrated Internal Handle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael D. April, Assistant Director for Research, Emergency Medicine Residency, Brooke Army Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: C.2015.046e
Record Dates: First submitted 2016-05-31; First posted 2016-06-07 (Estimated); Results first posted 2016-07-25 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-09

CONDITIONS: Apnea
MeSH Terms: conditions — Apnea

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Modified Ambu Spur II bag valve mask (Experimental): A health volunteer uses a modified Ambu Spur II bag valve mask with integrated internal handle (experimental device, not yet FDA approved) to deliver 10 breaths per minute for 3 minutes to a manikin (IngMar RespiTrainer manikin model).
  Interventions: Device: Modified Ambu Spur II bag valve mask
- Conventional Ambu Spur II bag valve mask (Active Comparator): A health volunteer uses a conventional Ambu Spur II bag valve mask to deliver 10 breaths per minute for 3 minutes to a manikin (IngMar RespiTrainer manikin model).
  Interventions: Device: Conventional Ambu Spur II bag valve mask

INTERVENTIONS:
Device: Modified Ambu Spur II bag valve mask — Subjects deliver breaths to manikin (IngMar RespiTrainer manikin model) a modified Ambu Spur II bag valve mask with integrated internal handle
  Arms: Modified Ambu Spur II bag valve mask
Device: Conventional Ambu Spur II bag valve mask — Subjects deliver breaths to manikin (IngMar RespiTrainer manikin model) a conventional Ambu Spur II bag valve mask
  Arms: Conventional Ambu Spur II bag valve mask

SUMMARY:
Investigators compared tidal volumes for single rescuer ventilation using a modified bag valve mask with an integrated internal handle versus a conventional bag valve mask in a manikin model.

DETAILED DESCRIPTION:
This was a prospective, randomized, crossover study to assess the tidal volume delivered using a standard and modified bag valve mask (BVM) device in a manikin airway model. Data was collected from July 2015 through October 2015 at the San Antonio Military Medical Center. Emergency medicine providers (physicians, physician assistants, residents, nurses, medics) were randomized to device order. Prior to participation each participant filled out a survey indicating their job status, gender, years of medical experience, and experience level with BVM ventilation. Hand grip strength and size (length, width, span) were measured. Each participant was then asked to provide BVM ventilation using the assigned devices at a rate of 10 breaths per minute for 3 minutes for a total of 30 breaths. Tidal volume of each delivered breath was recorded in milliliters. After a 3 minute rest period, testing was repeated with the second device. After ventilation with each device, participants completed an anonymous questionnaire that used a Likert scale to assess perceived qualities of the modified device including ease of use, ability to provide a superior mask seal, willingness to use in an emergency situation, and overall preference between the two devices. Each participant served as his/her own control.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Department healthy volunteers (physician assistants, residents, paramedics, nurses, medics, respiratory therapists.

Exclusion Criteria:

* Not trained in basic life support

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D April, MD, DPhil, Study Director — Brooke Army Medical Center
Locations (1):
- San Antonio Military Medical Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davidovic L, LaCovey D, Pitetti RD. Comparison of 1- versus 2-person bag-valve-mask techniques for manikin ventilation of infants and children. Ann Emerg Med. 2005 Jul;46(1):37-42. doi: 10.1016/j.annemergmed.2005.02.005. PMID 15988424
- [Background] Braude DA, Tawil I, Gerstein NS, Carey MC, Petersen TR. Comparison of bag-valve-mask hand-sealing techniques in a simulated model. Ann Emerg Med. 2014 Jun;63(6):784-5. doi: 10.1016/j.annemergmed.2014.01.037. No abstract available. PMID 24841402
- [Background] Otten D, Liao MM, Wolken R, Douglas IS, Mishra R, Kao A, Barrett W, Drasler E, Byyny RL, Haukoos JS. Comparison of bag-valve-mask hand-sealing techniques in a simulated model. Ann Emerg Med. 2014 Jan;63(1):6-12.e3. doi: 10.1016/j.annemergmed.2013.07.014. Epub 2013 Aug 9. PMID 23937957
- [Background] Amack AJ, Barber GA, Ng PC, Smith TB, April MD. Comparison of Ventilation With One-Handed Mask Seal With an Intraoral Mask Versus Conventional Cuffed Face Mask in a Cadaver Model: A Randomized Crossover Trial. Ann Emerg Med. 2017 Jan;69(1):12-17. doi: 10.1016/j.annemergmed.2016.04.017. Epub 2016 May 27. PMID 27238825

RESULTS

PARTICIPANT FLOW:
Groups:
- Modified Ambu Bag Valve Mask (BVM) First Then Unmodified BVM: A healthcare provider volunteer uses a modified Ambu Spur II bag valve mask with integrated internal handle (experimental device, not yet FDA approved) to deliver 10 breaths per minute for 3 minutes to a manikin (IngMar RespiTrainer manikin model). The subject then repeats these procedures using an unmodified Ambu bag valve mask.
- Unmodified Ambu Bag Valve Mask (BVM) First Then Modified BVM: A healthcare provider volunteer uses a conventional Ambu Spur II bag valve mask to deliver 10 breaths per minute for 3 minutes to a manikin (IngMar RespiTrainer manikin model). The subject then repeats these procedures using a modified Ambu Spur II bag valve mask with integrated handle.
Period: Overall Study
Arm/Group | Modified Ambu Bag Valve Mask (BVM) First Then Unmodified BVM | Unmodified Ambu Bag Valve Mask (BVM) First Then Modified BVM
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Modified Ambu Bag Valve Mask (BVM) First Then Unmodified BVM | Unmodified Ambu Bag Valve Mask (BVM) First Then Modified BVM | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 35 | 70
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 26 | 24 | 50
Region of Enrollment [Number; unit: participants]
  United States | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Mean Received Tidal Volume
Description: Each participant was asked to provide BVM ventilation using the assigned devices at a rate of 10 breaths per minute for 3 minutes for a total of 30 breaths. Tidal volume of each delivered breath was recorded in milliliters
Time Frame: 3 minutes
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | Modified Ambu Spur II Bag Valve Mask | Conventional Ambu Spur II Bag Valve Mask
Number analyzed (Participants) | 70 | 70
milliliters | 681 (148) | 591 (142)

2. Secondary Outcome: Modified Bag Valve Mask (BVM) Ease of Use
Description: Likert scale measuring subject's perceived ease of use of the modified BVM device from not at all easy to use (1) to very easy to use (5).
Time Frame: Within 10 minutes of study completion
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Modified Ambu Bag Valve Mask (BVM) First Then Unmodified BVM | Unmodified Ambu Bag Valve Mask (BVM) First Then Modified BVM
Number analyzed (Participants) | 35 | 35
Units on a scale | 5 [4 to 5] | 5 [4 to 5]

3. Secondary Outcome: Modified Bag Valve Mask (BVM) Better Seal Formation
Description: Subjects response using a Likert scale (1-5) regarding their perceptions of whether the modified BVM forms a better seal compared to a standard BVM: 1 (much worse seal formation) to 5 (much better seal formation).
Time Frame: Within 10 minutes of study completion
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Modified Ambu Bag Valve Mask (BVM) First Then Unmodified BVM | Unmodified Ambu Bag Valve Mask (BVM) First Then Modified BVM
Number analyzed (Participants) | 35 | 35
Units on a scale | 4 [3 to 4] | 4 [3 to 5]

4. Secondary Outcome: Modified Bag Valve Mask (BVM) Willingness to Use in Emergency Situation
Description: Subject reported willingness to use the modified BVM in a real life emergency situation as measured on a Likert scale ranging 1 (not at all willing to use) to 5 (very willing to use).
Time Frame: Within 10 minutes of study completion
Measure: Median (Inter-Quartile Range); unit: Units on a scale
Arm/Group | Modified Ambu Bag Valve Mask (BVM) First Then Unmodified BVM | Unmodified Ambu Bag Valve Mask (BVM) First Then Modified BVM
Number analyzed (Participants) | 35 | 35
Units on a scale | 5 [4 to 5] | 5 [4 to 5]

5. Secondary Outcome: Number of Participants Who Preferred the Modified Bag Valve Mask (BVM)
Description: Each subject provides a binary response as to whether he/she overall prefers using the modified BVM instead of the conventional BVM.
Time Frame: Within 10 minutes of study completion
Measure: Number; unit: participants
Arm/Group | Modified Ambu Bag Valve Mask (BVM) First Then Unmodified BVM | Unmodified Ambu Bag Valve Mask (BVM) First Then Modified BVM
Number analyzed (Participants) | 35 | 35
participants | 28 | 28

ADVERSE EVENTS:
Arm/Group | Modified Ambu Bag Valve Mask (BVM) First Then Unmodified BVM | Unmodified Ambu Bag Valve Mask (BVM) First Then Modified BVM
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No